CLINICAL TRIAL: NCT06344728
Title: A Phase 1, Open-Label, Randomized, Two-Period Crossover Study to Assess the Relative Bioavailability of Brensocatib Pediatric Oral Solution to Oral Tablets Following Single Oral Doses in Healthy Subjects
Brief Title: A Study to Assess the Relative Bioavailability of Brensocatib Pediatric Oral Solution to Oral Tablets in Healthy Participants
Acronym: INS1007
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: INS1007-110
Record Dates: First submitted 2024-03-27; First posted 2024-04-03 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Healthy Participants
MeSH Terms: interventions — brensocatib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Brensocatib Treatment Sequence AB (Experimental): Participants will receive a single dose of the pediatric oral brensocatib solution (Treatment A) on Day 1 followed by a washout period of 9 days. On Day 10, participants will receive a single dose of the oral brensocatib tablet (Treatment B).
  Interventions: Drug: Brensocatib Oral Solution; Drug: Brensocatib Oral Tablet
- Brensocatib Treatment Sequence BA (Experimental): Participants will receive a single dose of the oral brensocatib tablet (Treatment B) on Day 1 followed by a washout period of 9 days. On Day 10, participants will receive a single dose of the pediatric oral brensocatib solution (Treatment A).
  Interventions: Drug: Brensocatib Oral Solution; Drug: Brensocatib Oral Tablet

INTERVENTIONS:
Drug: Brensocatib Oral Solution — Brensocatib solution
  Other Names: INS1007
Drug: Brensocatib Oral Tablet — Brensocatib tablet
  Other Names: INS1007

SUMMARY:
The primary purpose of this study is to determine the relative bioavailability of brensocatib between the pediatric oral solution and oral tablets in healthy participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index between 18.0 and 32.0 kilogram per square meter (kg/m^2), and a body weight of ≥ 50 kilogram (kg) at Screening.
* Female participants of childbearing potential must have a negative urine or serum pregnancy test at Screening and Day -1 and agree to contraceptive requirements.
* To be a non-smoker and has not used chewing tobacco for at least 3 months prior to screening.
* Women must be postmenopausal (defined as no menses for 12 months without an alternative medical cause), surgically sterile, or using highly effective contraception from Screening to at least 30 days after discharge.
* Male participants must be on a stable method of contraception starting at Screening and continuing to at least 30 days after discharge.

Key Exclusion Criteria:

* History of stomach, gall bladder, or intestinal surgery or resection that would potentially alter absorption or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed).
* Administration of a coronavirus disease 2019 vaccine in the past 30 days prior to first dose.
* Use or intend to use any prescription medications/products other than hormone replacement therapy, oral, implantable, transdermal, injectable, or intrauterine contraceptives within 14 days prior to first dose.
* Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 60 days or 5 half-lives of that drug prior to first dose, whichever is longer.
* History of alcoholism or drug abuse within 2 years prior to check-in or 3 months before Screening, or excessive alcohol consumption (regular alcohol intake > 21 units per week for male participants and > 14 units of alcohol per week for female participants) (1 unit is equal to approximately 0.5 pint [200 milliliters (mL)] of beer, 1 small glass [100 mL] of wine, or 1 measure [25 mL] of spirits).
* Poor peripheral venous access. Note: Other inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Relative Bioavailability Between Brensocatib Pediatric Oral Solution and Oral Tablets for Area Under the Concentration-time Curve from Time 0 Extrapolated to Infinity (AUC∞) of Brensocatib in Plasma | Pre-dose and at multiple timepoints post-dose on Days 1 and 10
  Pharmacokinetics of brensocatib following a single dose in healthy participants will be assessed.

SECONDARY OUTCOMES:
Number of Participants who Experienced at Least one Adverse Event (AE) | Up to Day 23
Concentration of Brensocatib in Plasma | Pre-dose and at multiple timepoints post-dose on Days 1 and 10
  Pharmacokinetics of brensocatib following a single administration of different oral formulations in healthy participants will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- USA001, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No